## Chemotherapy Combined With Apatinib and PD-1 Monoclonal Antibody

## for Second-line or Above Treatment of Advanced Gastric Cancer

-A Prospective, Single-arm, Open, Phase II Study

Tianjin Medical University Cancer Hospital Informed Consent Version 1.0 (October 25, 2020)

The treatment of advanced gastric cancer is still dominated by chemotherapy. With the continuation of the treatment course, the sensitivity of advanced cancer patients to chemotherapy drugs will further decrease. In order to prolong the survival of such patients, second-line and post-line treatment is still needed. Irinotecan or taxanes can be selected for second-line treatment of advanced gastric cancer, but the effective rate of second-line chemotherapy is lower than 15%. However, for the third-line treatment of advanced gastric cancer, both the small-molecule targeted drug apatinib mesylate and the PD-1 antibody showed low single drug efficacy. Post-line treatment of advanced gastric cancer is difficult. Whether chemotherapy combined with immunization and targeting can be a new option for second-line or above treatment is a question worth exploring. Theoretically, chemotherapy can kill tumor cells and promote the release of tumor antigens, thus activating T cells and initiating immune circulation, so as to achieve synergistic effect with immunotherapy. The latest clinical results also show that first-line chemotherapy combined with immunotherapy has a survival benefit for advanced gastric cancer patients compared with chemotherapy alone. Apatinib mesylate is a targeted drug mainly anti-angiogenesis and PD-1 monoclonal antibody is an immunomodulator. Both of these drugs have been approved for the treatment of advanced gastric cancer. Preclinical studies have shown that PD-1 antibody and anti-angiogenic drugs can coordinate with each other to regulate tumor microenvironment, which is a very promising strategy for combined immunotherapy. A number of clinical studies have also confirmed that the combination of the two is safe and effective in the posterior line therapy of advanced gastric cancer. Based on the above theoretical basis, we believe that chemotherapy, immunotherapy and targeted anti-angiogenesis therapy have synergistic effects, which may achieve better anti-tumor effect and improve the effective rate of posterior line therapy for advanced gastric cancer patients. This study intends to give chemotherapy combined with PD-1 antibody and apatinib mesylate for advanced gastric cancer patients who need to receive second-line treatment or above. This three-drug regimen is expected to improve the effective rate of back-line treatment for advanced gastric cancer patients. You may have adverse reactions during the study. We will monitor all patients for any adverse reactions, and if you experience any adverse reactions between visits, please call your study physician immediately. The common adverse reactions of chemotherapy include bone marrow suppression (such as leukopenia,

neutrophil decline), gastrointestinal reactions (such as nausea, vomiting, diarrhea), etc. The common adverse reactions of apatinib include bone marrow suppression, proteinuria, hypertension, bleeding, gastrointestinal reactions and so on.Common adverse reactions of PD-1 monoclonal antibody include fatigue, hypothyroidism, immune hepatitis and so on. Clinically, these three drugs have good safety and controllable adverse reactions when used alone, but the risk of adverse reactions may increase when used in combination with the three drugs. For any adverse drug reactions that may occur during your participation in this study, the medical staff will closely observe the treatment process, actively give corresponding treatment measures, strictly grasp the application indications and termination conditions, and reduce accidents. Your participation in this study is voluntary, and you have the right to know the information related to you. Your privacy will be protected according to law, and your medical records will be kept confidential by the hospital and the client. Your medical records will become the study data of this drug, but your name will not be disclosed. If the results are published publicly in the journal, your identity will be kept confidential. This study was scientifically designed, followed the clinical application indications and instructions, and was approved by the Ethics Committee of the hospital. I have read the above content and understand the purpose of the study, as well as the possible advantages and disadvantages of participating in the study. The doctor in charge of the study has answered all my questions, and I voluntarily agree to participate in the clinical study.

| Patient Signature: | Date of signature: |
|-------------------------------------|--------------------|
| Signature of Witness (if required): | Date of signature: |
| Signature of Investigator: | Date of signature: |